CLINICAL TRIAL: NCT04834687
Title: Effects of Diet and Exercise Interventions on Cardiometabolic Risk Markers, Executive Function, and Intestinal Flora in Undergraduate Students: a Randomized Controlled Trial
Brief Title: Effects of Diet and Exercise Interventions on Cardiometabolic Risk Markers, Executive Function, and Intestinal Flora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanna Zhu, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZDGW[2021]044
Record Dates: First submitted 2021-04-03; First posted 2021-04-08 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Cardiometabolic Risk; Executive Function; Intestinal Microbiome
Keywords: Dietary Fiber; Time Restricted Feeding; Exercise; Young Adult
MeSH Terms: conditions — Intermittent Fasting; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rope-skipping group (Experimental): Participants would be required to take part in an exercise plan, under the instruction and guidance of professional sports teachers.
  Interventions: Behavioral: Exercise
- Diet intervention group (Experimental): Participants would be required to take part in a diet plan , including a high-fiber diet and time-restricted eating.
  Interventions: Behavioral: Diet
- Combined intervention group (Experimental): Participants will receive both rope-skipping and diet interventions at the same time.
  Interventions: Behavioral: Exercise; Behavioral: Diet
- Control group (No Intervention): Participants would be required to maintain existing diet patterns and physical activity levels.

INTERVENTIONS:
Behavioral: Exercise — Rope-skipping exercise for three times a week (90 minutes each time, and there is a 10 min break after 20 min Rope skipping). Exercise bracelet and smart bracelet would be used to record the energy consumption throughout the study.
  Arms: Combined intervention group; Rope-skipping group
Behavioral: Diet — Diet interventions include ten-hour time-restricted eating and a high-fiber diet.
  1. Participants will be instructed to take food from 7:30 AM until 5:30 PM and completely abstain from caloric intake for the remainder of the day (14 hours fast:10 hours eat). Only noncaloric beverages were permitted outside of the eating widow.
  2. According to the dietary recommendation proposed by Chinese Government and the existing dishes in the canteen , participants are instructed to eat following a high-diet recipe weekly from Monday to Friday which includes whole grain wheat rice, vegetables, fruits, and other foods rich in dietary fiber .
  Arms: Combined intervention group; Diet intervention group

SUMMARY:
The purpose of this study is to estimate the effects of diet and exercise interventions on body weight, cardiovascular metabolic markers, executive function, and intestinal flora among undergraduate students, as well as the underlying mechanisms.

DETAILED DESCRIPTION:
In recent decades, unhealthy dietary patterns and insufficiency of physical activity have brought negative effects on human health, such as rapid increasing incidence of obesity, metabolic cardiovascular diseases, and mental disorders. The first line of prevention and therapy for these diseases is proper diet and lifestyle interventions. A series of studies conducted in vivo and vitro have shown that high-fiber diets and time-restricted eating present benefits in weight loss, reducing cardiovascular disease risk, and improving cognitive function. While, there is also a randomized controlled trial do not observe the effects of time-restricted eating on weight loss and decrease of metabolic risks. Meanwhile, few studies have examined the effects of high-fiber diets or time-restricted eating on executive function. Additionally, previous studies on high-fiber diets and time-restricted eating focused on middle-aged or elderly populations with some features of metabolic syndrome, while the effects on healthy young populations are unclear. More importantly, there are a small amount of studies exploring the combined effects of time-restricted eating and physical activity on metabolism and cognitive function. Therefore, our study is to estimate the effects of diet (high-fiber diets and time-restricted eating) and exercise (rope-skipping) interventions on body weight, cardiovascular metabolic markers, executive function, and intestinal flora among undergraduate students, as well as the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* First and second year undergraduate students in Sun Yat-sen University.
* BMI≥22 kg/m^2.
* Keeping weight stable for 3 months prior to study start (weight fluctuation <5kg).
* Having the time and volunteering to receive the interventions.

Exclusion Criteria:

* Currently engaged in other weight-loss studies.
* With high blood pressure, diabetes or other cardiovascular diseases.
* With secondary obesity induced by medicine or other diseases.
* Contraindication to exercise.

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Body weight change of participants

SECONDARY OUTCOMES:
Body fat percentage | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Body fat percentage were measured by body composition analyzers.
Fat mass | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Fat mass (in kg) were measured by body composition analyzers.
Systolic and diastolic blood pressure | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Sitting systolic and diastolic blood pressure were measured with a validated electronic blood pressure monitor (model OMRON,HEM-7124).
Serum lipid levels | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Serum lipid levels (total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides) were analyzed by the enzymatic method.
Fasting plasma glucose | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Fasting plasma glucose were analyzed by the glucose oxidase method.
Fasting plasma insulin | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  Fasting plasma glucose were analyzed by the electrochemiluminescence method.
Intestinal flora | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  To measure the change of intestinal flora by analyzing feces genome 16S rDNA.
Change in scores on Behaviour Rating Inventory of Executive Functioning-Adult Version (BRIEF-A) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The executive functions were measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Self-Report Form. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Change in appetite sensations | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The appetite sensations were measured by the visual analogue scale (VAS).The VAS consisted of 100-mm lines and participants were required to place a vertical mark across the line corresponding best to their feelings of hunger, satisfaction, and fullness, with the scale ranging from 0 (not at all) to 100 (extremely). Quantification was performed by measuring the distance between the left end of the line and the vertical mark.
High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum hs-CRP were analyzed using the Luminex Human Magnetic Assay kit.
Intercellular adhesion molecule-1 (ICAM-1) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum ICAM-1 were analyzed using the Luminex Human Magnetic Assay kit.
Tumor necrosis factor alpha (TNF-alpha) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum TNF-alpha were analyzed using the Luminex Human Magnetic Assay kit.
Chemokine CCL2 | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum chemokine CCL2 were analyzed using the Luminex Human Magnetic Assay kit.
Vascular cell adhesion molecule (VCAM-1) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum VCAM-1 were analyzed using the Luminex Human Magnetic Assay kit.
Interleukin-6 (IL-6) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum IL-6 were analyzed using the Luminex Human Magnetic Assay kit.
Interleukin-8 (IL-8) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the IL-8 were analyzed using the Luminex Human Magnetic Assay kit.
Leptin | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum leptin were analyzed using the Luminex Human Magnetic Assay kit.
Tau protein | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum tau protein were analyzed using the Luminex Human Magnetic Assay kit.
Brain-derived neurotrophic factor (BDNF) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum BDNF were analyzed using the Luminex Human Magnetic Assay kit.
Vascular endothelial growth factor (VEGF) | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  The levels of the serum VEGF were analyzed using the Luminex Human Magnetic Assay kit.
Circulating metabolome | Baseline (1-2 days before the intervention), right after intervention (12 weeks)
  To measure the change of circulating metabolome by LC-MS/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: Yanna Zhu, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Maternal and Child Health and Sun Yat-sen Global Health Institute, School of Public Health and Institute of State Governance, Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Z, Li T, Huang F, Wu M, Zhu L, Zhou Y, Ming YA, Lu Z, Peng W, Gao F, Zhu Y. Comparison of diet and exercise on cardiometabolic factors in young adults with overweight/obesity: multiomics analysis and gut microbiota prediction, a randomized controlled trial. MedComm (2020). 2025 Jan 12;6(1):e70044. doi: 10.1002/mco2.70044. eCollection 2025 Jan. PMID 39802638
- [Derived] Lin Z, Zhang X, Wu M, Ming Y, Wang X, Li H, Huang F, Gao F, Zhu Y. High-fiber diet and rope-skipping benefit cardiometabolic health and modulate gut microbiota in young adults: A randomized controlled trial. Food Res Int. 2023 Nov;173(Pt 2):113421. doi: 10.1016/j.foodres.2023.113421. Epub 2023 Aug 30. PMID 37803759